CLINICAL TRIAL: NCT01890954
Title: Optimizing Closed-Loop Control of Type 1 Diabetes Mellitus in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16890
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Results first posted 2015-04-15 (Estimated); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes Mellitus (T1DM); Closed Loop Control (CLC); Diabetes Assistant (DiAs); Continuous Glucose Monitor (CGM)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DiAs-closed-loop system (Active Comparator): eight hours using Closed Loop Control (DiAs) under both, miss insulin bolus for 30 grams of carbohydrates snack or under bolus for an 80 grams of carbohydrates lunch
  Interventions: Device: Diabetes Assistant (DiAs)
- Sensor Augmented Pump (No Intervention): 8 hours observational under both, missed insulin bolus for 30 gr carbohydrates snack and under bolus for an 80 gr carbohydrates lunch. Sensor augmented pump used the patients own insulin settings (basal rate, meal boluses and correction boluses) and a CGM provided by the study team to be used during admission. No DiAs use during this admission.

INTERVENTIONS:
Device: Diabetes Assistant (DiAs) — Diabetes Assistance (DiAs) is a software residing in a Smartphone that contains the algorithms to regulate and control insulin deliveries (insulin bolus for: Basal rate, meal insulin and correction bolus) with inputs glucose values from a CGM and outputs insulin infusion by an insulin pump
  Other Names: Closed-Loop system
  Arms: DiAs-closed-loop system

SUMMARY:
The purpose of this study is to use a closed-loop Control-to-Range (CTR) system in adolescents with type 1 diabetes in an outpatient setting, and to evaluate the CTR system's ability to significantly improve blood glucose levels when an insulin bolus is omitted for a 30 gram carbohydrate snack and when insulin bolus is insufficient for the amount of carbohydrates consumed for a meal. The primary objective of this study is to use a closed-loop Control-to-Range (CTR) system to significantly reduce the post-prandial blood glucose excursion in adolescents with type 1 diabetes who omit and/or under-bolus insulin for either snacks or meals. Up to 20 subjects aged ≥13 and ≤18 years old will be tested.

DETAILED DESCRIPTION:
The purpose of this study is to use a closed-loop Control-to-Range (CTR) system in adolescents with type 1 diabetes in an outpatient setting, and to evaluate the CTR system's ability to significantly improve blood glucose levels when an insulin bolus is omitted for a 30 gram carbohydrate snack and when insulin bolus is insufficient for the amount of carbohydrates consumed for a meal. The CTR system is comprised of two algorithmic layers: (i) A Safety Supervision Module (SSM) which contains a predictive insulin request dampener (or brakes); (ii) a Range Correction Module (RCM), consisting in (a) a Hyperglycemia Mitigation System, and (b) Insulin on Board controller. Both modules will receive continuous glucose monitoring (CGM) and historical insulin delivery data. The SSM will monitor the safety of the subject's continuous subcutaneous insulin infusion pump (CSII) to prevent hypoglycemia. The RCM will be responsible for optimizing blood glucose (BG) control and mitigating postprandial hyperglycemic excursions through a mix of increased basal rate and, potentially, isolated insulin boluses. To run CTR, we will use our wearable artificial pancreas platform, known as DiAs (Diabetes Assistant) which consists of a smart phone running CTR and connected to standard insulin delivery and CGM devices.

ELIGIBILITY:
Inclusion Criteria:

1. ≥13 and ≤18 years old
2. Clinical diagnosis of type 1 diabetes mellitus for at least 2 years as noted by the following:

   Criteria for documented hyperglycemia (at least 1 criterion must be met):
   * Fasting glucose ≥126 mg/dL - confirmed
   * Two-hour Oral Glucose Tolerance Test (OGTT) ≥200 mg/dL - confirmed
   * Hemoglobin A1c (HbA1c) ≥6.5% documented by history - confirmed
   * Random glucose ≥200 mg/dL with symptoms
   * No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with diabetes

   Criteria for requiring insulin at diagnosis (at least 1 criterion must be met):
   * Participant required insulin at diagnosis and continually thereafter
   * Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually
   * Participant did not start insulin at diagnosis but continued to be hyperglycemic, had positive islet cell antibodies - consistent with Latent Autoimmune Diabetes in Adults (LADA) and did require insulin eventually and used continually
3. Use of an insulin pump to treat his/her diabetes for at least 6 months
4. Actively using a carbohydrate (CHO) /insulin ratio for insulin bolus adjustments in order to keep blood glucose in a predefined range
5. Tanner stage II or greater based on physician exam
6. HbA1c between <10.5% as measured with DCA2000 or equivalent device
7. Not currently known to be pregnant, breast feeding, or intending to become pregnant (females)
8. Demonstration of proper mental status and cognition for the study
9. Willingness to avoid consumption of acetaminophen-containing products during the study visits involving DexCom use
10. Self-reported behavior of snacking without insulin coverage or under bolus for meals
11. Willingness to consume a 30 grams snack without insulin coverage and willingness to bolus 75 % of usual treatment for an 80 grams lunch during both admissions
12. Willingness to remove home CGM for admissions if the subject typically wears a CGM
13. Medication stability in the preceding two months if taking antihypertensive, thyroid, anti-depressant or lipid lowering medication
14. Reported history of missed or inaccurate bolus treatments at meal time

Exclusion Criteria:

1. Diabetic ketoacidosis (DKA) within the 6 months prior to enrollment
2. In adherence with the One Touch Ultra 2 User Guide, subjects with hematocrit levels below 30% or above 55% will be excluded. Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
3. Pregnancy; breast feeding, or intention of becoming pregnant
4. Uncontrolled arterial hypertension (based on resting blood pressure > 95 percentile as listed according to age and height percentile in the Harriet Lane Handbook of Pediatrics)
5. Conditions which may increase the risk of hypoglycemia such as uncontrolled coronary artery disease during the previous year (e.g. history of myocardial infarction, acute coronary syndrome, therapeutic coronary intervention, coronary bypass or stenting procedure, stable or unstable angina, episode of chest pain of cardiac etiology with documented electrocardiogram (EKG) changes, or positive stress test or catheterization with coronary blockages >50%), congestive heart failure, history of cerebrovascular event, seizure disorder, syncope, adrenal insufficiency, neurologic disease or atrial fibrillation
6. History of a systemic or deep tissue infection with methicillin-resistant staph aureus or Candida albicans
7. History of arrythmia
8. Use of a device that may pose electromagnetic compatibility issues and/or radiofrequency interference with the DexCom CGM (implantable cardioverter-defibrillator, electronic pacemaker, neurostimulator, intrathecal pump, and cochlear implants)
9. Anticoagulant therapy other than aspirin
10. Oral steroids
11. Medical condition requiring use of an acetaminophen-containing medication that cannot be withheld for for 24 hours before CGM insertions until the end of each the study admissions.
12. Psychiatric disorders that would interfere with study tasks (e.g. inpatient psychiatric treatment within 6 months prior to enrollment)
13. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
14. Known current or recent alcohol or drug abuse
15. Medical conditions that would make operating a CGM, the DiAs cell phone, or insulin pump difficult (e.g. blindness, severe arthritis, immobility)
16. Any skin condition that prevents sensor or pump placement on the abdomen or arm (e.g. bad sunburn, pre-existing dermatitis, intertrigo, psoriasis, extensive scarring, cellulitis)
17. Impaired hepatic function measured as alanine aminotransferase or aspartate aminotransferase ≥ three times the upper reference limit
18. Impaired renal function measured as creatinine >1.2 times above the upper limit of normal
19. Uncontrolled microvascular (diabetic) complications (other than diabetic non-proliferative retinopathy), such as history of laser coagulation, proliferative diabetic retinopathy, known diabetic nephropathy (other than microalbuminuria with normal creatinine) or neuropathy requiring treatment
20. Active gastroparesis requiring current medical therapy
21. Uncontrolled thyroid disease
22. Known bleeding diathesis or dyscrasia
23. Known allergy to medical adhesives, components of the insulin pump insertion set or continuous glucose monitor sensor
24. Active enrollment in another clinical trial
25. Use of anti-diabetic agents other than continuous subcutaneous insulin infusion (CSII) including long-acting insulin, intermediate-acting insulin, metformin, sulfonylureas, meglitinides, thiazolidinediones, dipeptidyl peptidase 4 (DPP-4) inhibitors, glucagon-like peptide 1 agonists and alpha-glucosidase inhibitors
26. Subjects with basal rates less than 0.01 units/hour

RESTRICTIONS ON USE OF OTHER DRUGS OR TREATMENTS

1. Use of anti-diabetic agents other than CSII including long-acting insulin, intermediate-acting insulin, metformin, sulfonylureas, meglitinides, thiazolidinediones, DPP-4, inhibitors, glucagon-like peptide 1 agonists, and alpha-glucosidase inhibitors.
2. Acetaminophen will be restricted 24 hours before the insertion of not be allowed while the continuous glucose monitor is in use.
3. Medications that block symptoms of hypoglycemia, including but not limited to beta blockers.
4. Subjects on amylin analogs will be asked to withhold the medication during the outpatient admissions.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R. Chernavvsky, MD, CRC, Principal Investigator — University of Virginia; Mark DeBoer, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make de-identified individual participant data (IPD) collected in this study available to other researchers at the end of the study. Paper published in Pediatric Diabetes

REFERENCES:
- [Result] Chernavvsky DR, DeBoer MD, Keith-Hynes P, Mize B, McElwee M, Demartini S, Dunsmore SF, Wakeman C, Kovatchev BP, Breton MD. Use of an artificial pancreas among adolescents for a missed snack bolus and an underestimated meal bolus. Pediatr Diabetes. 2016 Feb;17(1):28-35. doi: 10.1111/pedi.12230. Epub 2014 Oct 27. PMID 25348683

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care First, Then Closed Loop Control: 8 hours observational (09:00-17:00) during usual care with a missed insulin bolus for 30g carbohydrates snack (09:00) and an under-bolus (75% meal insulin with full correction insulin) for an 80g lunch (13:00). 1 day of wash-out. 8 hours using Closed Loop Control with DiAs with a missed insulin bolus for 30g of carbohydrates snack (09:00) and an under-bolus (75% meal insulin with no correction insulin) for an 80g lunch (13:00).
- Closed Loop Control First, Then Usual Care: 8 hours observational (09:00-17:00) using Closed Loop Control with DiAs with a missed insulin bolus for 30g of carbohydrates snack (09:00) and an under-bolus (75% meal insulin with no correction insulin) for an 80g lunch (13:00). 1 day of wash-out. 8 hours observational (09:00-17:00) during usual care with a missed insulin bolus for 30g carbohydrates snack (09:00) and an under-bolus (75% meal insulin with full correction insulin) for an 80g lunch (13:00).
Period: Overall Study
Arm/Group | Usual Care First, Then Closed Loop Control | Closed Loop Control First, Then Usual Care
Started | 9 | 8
Completed | 8 | 8
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Closed Loop Control First, Then Usual Care: 8 hours observational (09:00-17:00) using Closed Loop Control with DiAs with a missed insulin bolus for 30g of carbohydrates snack (09:00) and an under-bolus (75% meal insulin with no correction insulin) for an 80g lunch (13:00). 1 day of wash-out. 8 hours observational during usual care with a missed insulin bolus for 30g carbohydrates snack (09:00) and an under-bolus (75% meal insulin with full correction insulin) for an 80g lunch (13:00).
- Total: Total of all reporting groups
Arm/Group | Usual Care First, Then Closed Loop Control | Closed Loop Control First, Then Usual Care | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 8 | 16
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (2) | 15 (2) | 15 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percent of Time Spent Near Normoglycemia
Description: Percentage of time that blood glucose (BG) values (measured with both finger-stick and CGM) were near normoglycemia (70-180 mg/dL).
Time Frame: 8 hours
Measure: Mean (Standard Error); unit: percentage time near normoglycemia
Groups:
- Closed Loop Control With DiAs System: 8 hours observational (09:00-17:00) during closed-loop control (DiAs) with a missed insulin bolus for 30g carbohydrates snack (09:00) and an under-bolus (75% meal insulin with full correction insulin) for an 80g lunch (13:00).
- Usual Care Without DiAs System (CGM Only): 8 hours observational (09:00-17:00) during usual care with a missed insulin bolus for 30g carbohydrates snack (09:00) and an under-bolus (75% meal insulin with full correction insulin) for an 80g lunch (13:00).
Arm/Group | Closed Loop Control With DiAs System | Usual Care Without DiAs System (CGM Only)
Number analyzed (Participants) | 16 | 16
percentage time near normoglycemia
  Overall (8 hours) | 43.4 (6.5) | 18.9 (7)
  Post-snack (4 hours) | 45.1 (8.7) | 21.3 (7.7)
  Post-lunch (4 hours) | 42.3 (9.2) | 16.9 (7.4)

ADVERSE EVENTS:
Groups:
- Closed Loop Control With DiAs System: 8 hours using Closed Loop Control with DiAs under both, miss insulin bolus for 30 grams of carbohydrates snack or under bolus for an 80 grams of carbohydrates lunch
  Diabetes Assistant (DiAs)
- Usual Care Without DiAs System (CGM Only): 8 hours observational under both, missed insulin bolus for 30 gr carbohydrates snack and under bolus for an 80 gr carbohydrates lunch.
Arm/Group | Closed Loop Control With DiAs System | Usual Care Without DiAs System (CGM Only)
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
BG values followed 4 h after the unannounced meals, risk for hypoglycemia could have been detected if followed longer

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes